CLINICAL TRIAL: NCT01606358
Title: IClyCO Influence of Chemotherapy (Carboplatin and Taxol) on the ex Vivo Expansion and Functional Capacity of Gamma-delta T Cells in Patients With Epithelial Ovarian Cancer
Brief Title: Influence of Chemotherapy on Gamma-delta T Cells in Patients With Epithelial Ovarian Cancer
Acronym: IClyCO
Status: Withdrawn | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00214-37
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Patient with ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The VGAMMA9VDELTA2 T cells will be isolated from peripheral blood mononuclear cells of patients with ovarian cancer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian Cancer
  Interventions: Drug: Carboplatin and / or taxol chemotherapy

INTERVENTIONS:
Drug: Carboplatin and / or taxol chemotherapy — Patient with proven epithelial ovarian cancer and receiving carboplatin and / or taxol chemotherapy (usual care).

SUMMARY:
In patients with an ovarian cancer, the treatment is currently based on surgery and chemotherapy.

The impact of chemotherapy on the expansion and functional abilities of Vgamma9Vdelta2 T cells has never been evaluated.

The long term goal is to give a rational to combine conventional treatment of ovarian cancer with immunotherapy based on Vgamma9Vdelta2 T cells.

DETAILED DESCRIPTION:
Ovarian cancer is associated with a high mortality rate. Treatment of ovarian cancer is currently based on surgery and chemotherapy.

The first surgery is a radical surgical procedure aiming to achieve no residual disease. Patients who could not benefit from the first surgery may be offered neoadjuvant chemotherapy with a new surgical procedure after 3 or 6 chemotherapy cycles. Chemotherapy is currently based on Taxol and Carboplatin. Immunotherapy based on Vgamma9Vdelta2 T cells could provide a promising therapeutic strategy, however, the impact of chemotherapy on the expansion and functional abilities of Vgamma9Vdelta2 T cells has never been evaluated.

We want to study the effect of chemotherapy of ovarian cancer on Vgamma9Vdelta2 T cells rates in the peripheral blood of patients with ovarian cancer.

Functional abilities of the Vgamma9Vdelta2 T cells will be studied: expansion after chemotherapy and their cytotoxic abilities in an autologous context before or after chemotherapy.

The long term goal is to give a rational to combine conventional treatment of ovarian cancer with non-conventional treatment such as immunotherapy based on Vgamma9Vdelta2 T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven epithelial ovarian cancer
* Patients receiving carboplatin and / or taxol chemotherapy.

Exclusion Criteria:

* Minor patient
* Protected adult
* Lack of invasion to the final histological checking
* Absence of chemotherapy in the therapeutic plan of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with proven epithelial ovarian cancer and receiving carboplatin and / or taxol chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD PhD, Study Chair — Rennes University Hospital
Locations (1):
- CHU de RENNES, Rennes, France